CLINICAL TRIAL: NCT03460405
Title: Safety and Immunogenicity of Vi-DT Typhoid Conjugate Vaccine (Bio Farma) in Indonesian Adults, Adolescents, Children and Infants (Phase II)
Brief Title: Safety and Immunogenicity of Vi-DT Typhoid Conjugate Vaccine in Indonesian Adults, Adolescents, Children and Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Typhoid 0218
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Safety Issues; Immunogenicity
MeSH Terms: interventions — Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Intervention Model Description: Subject aged 2 - 40 years old:
  Randomized, observer-blind, superiority design compared to Vi polysaccharide vaccine.
  Subject aged 6-23 months old:
  Randomized, observer-blind, superiority design compared to Inactivated Poliomyelitis Vaccine (IPV).
Who Masked: Participant, Investigator
Masking Description: Subject aged 2 - 40 years old:
  Randomized, observer-blind, superiority design compared to Vi polysaccharide vaccine.
  Subject 6-23 months old:
  Randomized, observer-blind, superiority design compared to Inactivated Poliomyelitis Vaccine (IPV).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- VI-DT vaccine (adults,adolescent) (Experimental): 1 dose of 0.5 ml Vi-DT vaccine
  Interventions: Biological: Vi-DT Vaccine
- Vi polysaccharide (adults,adolescent) (Active Comparator): 1 dose of 0.5 ml Vi polysaccharide vaccine
  Interventions: Biological: Vi Polysaccharide Vaccine
- VI-DT vaccine (children) (Experimental): 1 dose of 0.5 ml Vi-DT vaccine
  Interventions: Biological: Vi-DT Vaccine
- Vi polysaccharide vaccine (children) (Active Comparator): 1 dose of 0.5 ml Vi polysaccharide vaccine
  Interventions: Biological: Vi Polysaccharide Vaccine
- VI-DT vaccine (infants) (Experimental): 1 dose of 0.5 ml Vi-DT vaccine
  Interventions: Biological: Vi-DT Vaccine
- IPV Vaccine (infants) (Active Comparator): 1 dose of 0.5 ml IPV vaccine
  Interventions: Biological: IPV Vaccine

INTERVENTIONS:
Biological: Vi-DT Vaccine — 1 dose of Vi-DT Vaccine
  Other Names: Typhoid Conjugate Vaccine
  Arms: VI-DT vaccine (adults,adolescent); VI-DT vaccine (children); VI-DT vaccine (infants)
Biological: Vi Polysaccharide Vaccine — 1 dose of Vi Polysaccharide Vaccine
  Arms: Vi polysaccharide (adults,adolescent); Vi polysaccharide vaccine (children)
Biological: IPV Vaccine — 1 dose of IPV Vaccine
  Arms: IPV Vaccine (infants)

SUMMARY:
This study is to assess the safety and immunogenicity of Vi-DT vaccine in adults, adolescent, children and infants.

DETAILED DESCRIPTION:
To describe the safety of this vaccine following one dose immunization in adults, adolescent, children and infants.

To assess immunogenicity following one dose of Vi-DT vaccine immunization. To compare the safety and immunogenicity of Vi-DT to Vi polysaccharide vaccine in adults, adolescents, and children groups.

To compare the safety and immunogenicity of Vi-DT to IPV vaccine in infants groups.

Kinetics of Vi-specific IgG antibodies up to 6 months and 1 year after administration of 1 dose of vaccine.

To evaluate the safety and immunogenicity of Vi-DT co-administered with MR vaccine in infants (≥ 9months -23 months old).

To evaluate the safety and immunogenicity of MR vaccine co-administered with Vi-DT vaccine in infants (≥ 9months -23 months old).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy
2. Subjects/Parents have been informed properly regarding the study and signed the informed consent form
3. Subject/parents/legal guardians will commit themselves to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria For adults-adolescent-children:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial
2. Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature ³ 37.5°C)
3. Known history of allergy to any component of the vaccines
4. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
5. Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products, corticosteroid therapy and other immunosuppresant).
6. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives
7. Pregnancy & lactation (Adults)
8. Individuals who have previously received any vaccines against typhoid fever.
9. Subjects already immunized with any vaccine within 1 month prior and expect to receive other vaccines within 1 month following immunization.
10. Individuals who have a previously ascertained typhoid fever within 3 months prior to immunization.
11. History of substance abuse (Adults).
12. Subject planning to move from the study area before the end of study period.

Exclusion Criteria for infants:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial
2. Mother less than 18 years of age at the age of enrollment of the infant
3. Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature ³ 37.5°C)
4. Known history of allergy to any component of the vaccines
5. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
6. Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products, corticosteroid therapy and other immunosuppresant).
7. Any abnormality or chronic disease which according to the investigator might be compromised by the vaccination and/or interfere with the assessment of the trial objectives.
8. Individuals who have previously received any vaccines against typhoid fever.
9. Subjects already immunized with any vaccine within 1 month prior and expect to receive other vaccines within 1 month following immunization, except MR vaccine.
10. Individuals who have a previously ascertained typhoid fever within 3 months prior to immunization.
11. Subject planning to move from the study area before the end of study period.

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Local reaction and systemic event after vaccination | 28 days
  Percentage of subjects with at least one immediate reaction (local reaction or systemic event) after vaccination.

SECONDARY OUTCOMES:
Adverse events after vaccination | up to 28 days
  Percentage of subjects with at least one of these adverse events, solicited or not, within 24 h, 48h, 72h and 28 days after 1 dose vaccination.
Serious adverse events after vaccination | 28 days
  Number and percentage of subjects with serious adverse event from inclusion until 28 day after vaccination
Geometric Mean Titers (GMT) | 28 days
  Geometric Mean Titers (GMT) 28 days following immunization
Percentage of subjects with increasing antibody titer >= 4 times | 28 days
  Percentage of subjects with increasing antibody titer >= 4 times in all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Bernie Endyarni, MD, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (2):
- Indonesia (2):
  - Puskesmas Jatinegara, Jakarta
  - Puskesmas Senen, Jakarta

REFERENCES:
- [Derived] Koesnoe S, Medise BE, Rengganis I, Hadinegoro SR, Puspita M, Sari RM, Yang JS, Sahastrabuddhe S, Soedjatmiko, Gunardi H, Sekartini R, Wirahmadi A, Kekalih A, Mukhi S, Satari HI, Bachtiar NS. A phase II clinical trial of a Vi-DT typhoid conjugate vaccine in healthy Indonesian adolescents and adults: one-month evaluation of safety and immunogenicity. Trop Dis Travel Med Vaccines. 2024 Feb 1;10(1):3. doi: 10.1186/s40794-023-00210-z. PMID 38297337
- [Derived] Medise BE, Soedjatmiko S, Gunardi H, Sekartini R, Satari HI, Hadinegoro SR, Wirahmadi A, Puspita M, Sari RM, Yang JS, Sil A, Sahastrabuddhe S, Bachtiar NS. A novel Vi-diphtheria toxoid typhoid conjugate vaccine is safe and can induce immunogenicity in healthy Indonesian children 2-11 years: a phase II preliminary report. BMC Pediatr. 2020 Oct 15;20(1):480. doi: 10.1186/s12887-020-02375-4. PMID 33059607
- [Derived] Medise BE, Soedjatmiko S, Gunardi H, Sekartini R, Satari HI, Hadinegoro SR, Wirahmadi A, Puspita M, Sari RM, Yang JS, Sil A, Sahastrabuddhe S, Bachtiar NS. One-month follow up of a randomized clinical trial-phase II study in 6 to <24 months old Indonesian subjects: Safety and immunogenicity of Vi-DT Typhoid Conjugate Vaccine. Int J Infect Dis. 2020 Apr;93:102-107. doi: 10.1016/j.ijid.2020.01.045. Epub 2020 Jan 28. PMID 32004693